CLINICAL TRIAL: NCT02502630
Title: CT-guided Percutaneous Microwave Ablation for Pulmonary Metastases From Colorectal Cancer
Brief Title: Microwave Ablation for Pulmonary Metastases From Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-MW-001
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated with microwave ablation (Experimental): Patients undergoing MWA for pulmonary metastases from colorectal cancer.
  Interventions: Device: microwave ablation

INTERVENTIONS:
Device: microwave ablation — pulmonary metastases from colorectal cancer are destructed/ablated using microwave ablation

SUMMARY:
(MWA) is the most recent development in the field of local ablative therapies. The aim of this study was to evaluate CT-guided percutaneous microwave (MW) ablation safety and efficacy in pulmonary metastases from colorectal cancer.

DETAILED DESCRIPTION:
From June 2010 to June 2015, 48 unresectable lesions in 32 patients with pulmonary metastases from colorectal cancer were selected for CT-guided microwave ablation. Patients were scheduled for a 1 and 3 month CT follow-up to evaluate lesion diameter.We retrospectively evaluated CT-guided percutaneous microwave (MW) ablation safety and efficacy in pulmonary metastases from colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable pulmonary metastases from colorectal cancer.
* diagnosis by CT, and confirmed by percutaneous puncture biopsy.
* Age range 18-70 years old.
* Eastern Cooperative Oncology Group performance status 0-1.
* Life expectancy of more than 3 months.
* Adequate organ function.

Exclusion Criteria:

* Resectable lung metastases.
* Life expectancy less than 3 months
* Patients with cardiac pacemaker, cerebral aneurysm clips, implanted electronic instruments or other metal materials.
* Coagulopathy with platelet count less than 50000.
* Active infectious disease.
* Age below 18 years.
* Pregnancy of breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | one year

SECONDARY OUTCOMES:
Treatment related adverse events | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jingting Jiang, PD, Study Director — The First People's Hospital of Changzhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cheng G, Shi L, Qiang W, Wu J, Ji M, Lu Q, Li X, Xu B, Jiang J, Wu C. The safety and efficacy of microwave ablation for the treatment of CRC pulmonary metastases. Int J Hyperthermia. 2018 Jun;34(4):486-491. doi: 10.1080/02656736.2017.1366553. Epub 2017 Nov 16. PMID 28847194